CLINICAL TRIAL: NCT06012864
Title: Modified Flank-free Supine Versus Prone PNL in Pediatric Renal Stones: A Prospective Randomized Comparative Trial
Brief Title: Supine Versus Prone PNL in Pediatric
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Kamel Abdel Rahman, DR, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Supine pediatric PNL
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: Patients divided into two groups (group A: modified supine PNL, group B: prone PNL)
Who Masked: Participant
Masking Description: closed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified supine PNL (Experimental): patients doing FFMS PNL
  Interventions: Procedure: PNL
- prone PNL (Experimental): patients doing prone PNL
  Interventions: Procedure: PNL

INTERVENTIONS:
Procedure: PNL — percutaneous extraction of the stones in the kidney

SUMMARY:
To Compare the safety and efficacy of PNL in a modified flank-free supine position versus prone position in pediatric patients

DETAILED DESCRIPTION:
Incidence of pediatric urolithiasis varies from 5%-15% in developing countries to 1%-5% in the developed ones. The 5-year recurrence rate of about55% (range, 38%-70%). Fernstrom and Johansson first introduced percutaneous nephrolithotomy (PNL) in 1976. Since that PNL has become widely used for multiple indications. Pediatric PNL was done in the prone position with more rapid and easy puncture point determination, wider field for renal puncture, free application of multiple accesses, and avoidance of visceral injuries, especially the colon. PNL in the supine position has several advantages as, similar success rate and a shorter operative time than conventional PNL. The Amplatz sheath is oriented downward, maintaining a low pressure in the renal pelvis and reducing the fluid absorption with rapid drainage of the fragmented stones. Furthermore, it's easier for the anesthesiologist to control the airway and reduce the neural and ophthalmologic pressure lesions than the prone position. Desoky et al in 2012 described the flank-free modified supine position (FFMSP) and claimed that this position overcomes the mechanical limitation of ordinary supine position because of ample space for puncture, dilatation, multiple tracts, and maneuverability of the system with the nephoscope. Moreover, the surgeon can comfortably sit during the operation, and X-ray exposure is reduced because puncture and dilatation are quite perpendicular to the body, and the operator's hands are outside the fluoroscopic field. it's better to do supine PNL in case of retro renal colon. as we see the supine position in pediatric is still under research and few trials about it had been done with no clear recommendation, so we will compare PNL in pediatric age group in modified free flank supine position versus prone position.

ELIGIBILITY:
Inclusion Criteria:

Age ≤ 18 years old. Renal stones are amenable for PNL with Guy's stone score 1-2.

Exclusion Criteria:

congenital anomalies. skeletal anomalies. bleeding diathesis. active urinary tract infection. Patient refusing participation. Patients with PCN.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
sucess rate | within 3 months post operative
  stone free rate

SECONDARY OUTCOMES:
complication rate | 1 month
  rate of patients develop complication
operative time | intraoperative
  from the puncture untill the end

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Eltaher, MD, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holman E, Khan AM, Flasko T, Toth C, Salah MA. Endoscopic management of pediatric urolithiasis in a developing country. Urology. 2004 Jan;63(1):159-62; discussion 162. doi: 10.1016/j.urology.2003.08.043. PMID 14751372
- [Background] Lao M, Kogan BA, White MD, Feustel PJ. High recurrence rate at 5-year followup in children after upper urinary tract stone surgery. J Urol. 2014 Feb;191(2):440-4. doi: 10.1016/j.juro.2013.09.021. Epub 2013 Sep 16. PMID 24050895
- [Background] Liatsikos EN, Kallidonis P, Stolzenburg JU, Ost M, Keeley F, Traxer O, Bernardo N, Perimenis P, Smith AD. Percutaneous management of staghorn calculi in horseshoe kidneys: a multi-institutional experience. J Endourol. 2010 Apr;24(4):531-6. doi: 10.1089/end.2009.0264. PMID 20218888
- [Background] Caione P, De Dominicis M, Collura G, Matarazzo E, Nappo SG, Capozza N. Microperc for pediatric nephrolithiasis: technique in valdivia-modified position. Eur J Pediatr Surg. 2015 Feb;25(1):94-9. doi: 10.1055/s-0034-1387939. Epub 2014 Sep 13. PMID 25217714
- [Background] Desoky EAE, Sakr AM, ElSayed ER, Ali MM. Ultra-Mini-Percutaneous Nephrolithotomy in Flank-Free Modified Supine Position vs Prone Position in Treatment of Pediatric Renal Pelvic and Lower Caliceal Stones. J Endourol. 2022 May;36(5):610-614. doi: 10.1089/end.2021.0557. Epub 2022 Mar 9. PMID 34861776
- [Background] Falahatkar S, Moghaddam AA, Salehi M, Nikpour S, Esmaili F, Khaki N. Complete supine percutaneous nephrolithotripsy comparison with the prone standard technique. J Endourol. 2008 Nov;22(11):2513-7. doi: 10.1089/end.2008.0463. PMID 19046091
- [Background] Vicentini FC, Torricelli FC, Mazzucchi E, Hisano M, Murta CB, Danilovic A, Claro JF, Srougi M. Modified complete supine percutaneous nephrolithotomy: solving some problems. J Endourol. 2013 Jul;27(7):845-9. doi: 10.1089/end.2012.0725. Epub 2013 Jun 8. PMID 23373958
- [Background] Kukreja RA, Desai MR, Sabnis RB, Patel SH. Fluid absorption during percutaneous nephrolithotomy: does it matter? J Endourol. 2002 May;16(4):221-4. doi: 10.1089/089277902753752160. PMID 12042103
- [Background] Desoky EA, Allam MN, Ammar MK, Abdelwahab KM, Elsaid DA, Fawzi AM, Alayman AA, Shahin AM, Kamel HM. Flank free modified supine position: A new modification for supine percutaneous nephrolithotomy. Arab J Urol. 2012 Jun;10(2):143-8. doi: 10.1016/j.aju.2011.12.008. Epub 2012 Mar 7. PMID 26558017
- [Background] De Sio M, Autorino R, Quarto G, Calabro F, Damiano R, Giugliano F, Mordente S, D'Armiento M. Modified supine versus prone position in percutaneous nephrolithotomy for renal stones treatable with a single percutaneous access: a prospective randomized trial. Eur Urol. 2008 Jul;54(1):196-202. doi: 10.1016/j.eururo.2008.01.067. Epub 2008 Feb 4. PMID 18262711
- [Background] Emiliani E, Quiroz YY, Llorens E, Quintian C, Motta G, Villada D, Bujons A. Retrorenal colon in pediatric patients with urolithiasis: Is the supine position for PCNL advantageous? J Pediatr Urol. 2022 Dec;18(6):741.e1-741.e6. doi: 10.1016/j.jpurol.2022.07.028. Epub 2022 Aug 3. PMID 35985922